CLINICAL TRIAL: NCT06602947
Title: To Compare the Consumption of Sevoflurane and Desflurane in Low-flow Anesthesia Using the Recommendations of ASA (American Society of Anaesthesiologist Environmental Sustainability Committee
Brief Title: To Compare the Consumption of Sevoflurane and Desflurane in Low Flow Anaesthesia
Status: Completed | Type: Observational
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr soumi pathak, Consultant Anaesthesia, Rajiv Gandhi Cancer Institute & Research Center, India
Other Study IDs: Res/SCM/23/2017/53
Record Dates: First submitted 2021-09-19; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Sevoflurane; Desflurane
Keywords: Low flow anesthesia; carbon footprint

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low-flow sevoflurane (LFS): Anaesthesia will be administered according to the recommendations of ASA Enviornment Sustainability Committee.
  Three strategies to reduce the fresh gas flow and enviornmental contamination are
  1. Induction: Set the Vaporizer to Deliver a Concentration Greater than Intended
  2. Intubation: Turn Off the Fresh Gas Flow, Not the Vaporizer.
  3. Maintanance: Minimize Fresh Gas Flow During Maintenance.
  Interventions: Other: Low flow anaesthesia using ASA enviormental sustanibility commitee recomendation
- low- flow desflurane (LFD): Anaesthesia will be administered according to the recommendations of ASA Enviornment Sustainability Committee.
  Three strategies to reduce the fresh gas flow and enviornmental contamination are
  1. Induction: Set the Vaporizer to Deliver a Concentration Greater than Intended
  2. Intubation: Turn Off the Fresh Gas Flow, Not the Vaporizer.
  3. Maintanance: Minimize Fresh Gas Flow During Maintenance.
  Interventions: Other: Low flow anaesthesia using ASA enviormental sustanibility commitee recomendation

INTERVENTIONS:
Other: Low flow anaesthesia using ASA enviormental sustanibility commitee recomendation — 1. Induction: Set the Vaporizer to Deliver a Concentration Greater than Intended
  2. Intubation: Turn Off the Fresh Gas Flow, Not the Vaporizer.
  3. Maintanance: Minimize Fresh Gas Flow During Maintenance.

SUMMARY:
This prospective observational study aims to compare sevoflurane and Desflurane consumption in low-flow anaesthesia using the ASA (American Society of Anaesthesiology).

Environmental Sustainability Committee recommendations. The patients aged 20-65 years, ASA I and II undergoing surgery under general anaesthesia were included in the study.

Question: Can we reduce our carbon footprint of desflurane and sevoflurane using low-flow anaesthesia, according to the recommendations of the ASA Environment Sustainability Committee?

PRIMARY To compare the mac hour consumption of sevoflurane and desflurane anaesthetic agents under low flow (one litre/min) conditions To calculate the carbon footprint of sevoflurane and desflurane in the study cases.

SECONDARY To test whether a significant generation of carbon monoxide occurs due to the interaction of sevoflurane/desflurane with soda lime in the closed circuit Groups 1) low-flow sevoflurane (LFS)- 1 L/min gas flow 2) low- flow desflurane (LFD)- 1 L/min gas flow Anaesthesia will be administered according to the recommendations of the ASA Environment Sustainability Committee.

Three strategies to reduce the fresh gas flow and environmental contamination are

1. Induction: Set the Vaporizer to Deliver a Concentration Greater than Intended
2. Intubation: Turn Off the Fresh Gas Flow, Not the Vaporizer.
3. Maintenance: Minimize Fresh Gas Flow During Maintenance.

DETAILED DESCRIPTION:
OBJECTIVES

PRIMARY To compare the mac hour consumption of sevoflurane and desflurane anaesthetic agents under low flow (one litre/min) conditions To calculate the carbon footprint of sevoflurane and desflurane in the low-flow anaesthesia being used in this study

SECONDARY To test whether a significant generation of carbon monoxide occurs due to the interaction of sevoflurane/desflurane with soda lime in the closed circuit.

Methodology Two groups: 1) low-flow sevoflurane (LFS) 2) low- flow desflurane (LFD) Anaesthesia will be administered according to the recommendations of the ASA Environment Sustainability Committee.

Three strategies to reduce the fresh gas flow and environmental contamination are

1. Induction: Set the Vaporizer to Deliver a Concentration Greater than Intended
2. Intubation: Turn Off the Fresh Gas Flow, Not the Vaporizer.
3. Maintenance: Minimize Fresh Gas Flow During Maintenance.

Five hundred sixty-four patients aged 20-65 and ASA status I-II scheduled for procedures longer than three hours duration at Rajiv Gandhi Cancer Institute & Research Center (RGCI&RC) from 2017-2018 will be included in this study.

Patients having severe cardiac and hepatic problems, renal dysfunction and chronic alcoholism are excluded from the study Computer-generated randomisation will be done to allocate the patients into two equal groups for low-flow sevoflurane and low-flow desflurane anaesthesia.

After the arrival of the patients, aVenous cannula will be inserted; midazolam 0.05 mg. kg-1 will be administered intravenously for anxiolysis. Noninvasive monitors, including electrocardiograms, non-invasive blood pressure monitoring, pulse oximetry, axillary temperature, and bispectral index (BIS), will be applied.

Anaesthesia will be induced with fentanyl (2µg.kg-1 ), propofol (2.5 mg. kg-1 ) and atracurium (0.5mg. kg -1 ) to facilitate endotracheal intubation.

All patients will be mechanically ventilated with a mixture of air-oxygen (50% oxygen + 50% air) in addition to the anaesthetic agent according to the study group using the anaesthesia workstation (Primus®, Dräger, Luebeck, Germany).

The tidal volume will be set at 8mL/kg, and the respiratory frequency will be to maintain an end-tidal CO 2 (Et CO2 ) between 30-35mmHg.

After intubation, anaesthesia will be maintained with the fresh gas flow (FRF) of 4 lit./min and 4% Vol sevoflurane or 6% Vol desflurane in the 50% oxygen/air mixture for 5 minutes.

The fresh gas flow will be decreased to 1 L min-1, and after that, dial concentration will be reduced by 0.5% every 2 minutes to maintain 1 MAC(minimum alveolar concentration).

The dial concentration after that will be adjusted to achieve a value of 1 MAC. An adequate neuromuscular blockade will be achieved by administering atracurium boluses of 0.1mg. kg-1 every 20min.

During skin closure, the anaesthetic will be discontinued, and the patient will receive 100% O 2.

At 25% recovery of the first response to train-of-four stimulation, the neuromuscular blockade will be reversed by neostigmine (4µg.kg-1 ) and atropine (15µg.kg-1 ). ABG( Arterial blood gas) were done baseline and post-procedure.

PARAMETERS TO BE RECORDED:

A. Carbon footprint calculation.

1. Consumption of the anaesthetic agent will be recorded from the logbook Draeger Primus™ on termination of anaesthesia
2. Consumed inhalational agent (ml) in 1 MAC hour. Consumption of the inhalational agent (ml) will be converted to MAC hour consumption by dividing it by the entire duration of 1.0 MAC anaesthesia.
3. Calculation of carbon dioxide equivalent. The consumed inhalational agent (ml) will be converted to tones by volume weight conversion formula (1.465 for Desflurane and 1.522 for Sevoflurane) and then multiplied by( Global warming potential) GWP100 (2540 for Desflurane and 130 for Sevoflurane) to get carbon dioxide equivalent.
4. Estimation of carboxy haemoglobin (CoHb) levels as read from ABG analysis on termination of anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with American Society of Anesthesiologists grade (ASA) I & II.
2. Patients with age 20-65 years.

Exclusion Criteria:

1. Contraindications to inhalation agents.
2. Liver dysfunction.
3. Chronic alcoholism.
4. Chronic smokers.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 564 patients aged 20-65 and ASA status I-II scheduled for procedures longer than three hours duration at RGCI&RC from 2017-2018 will be included in this study
Sampling Method: Probability Sample
Enrollment: 564 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
To compare the MAC hour consumption of sevoflurane under low flow conditions. To compare the mac hour consumption of sevoflurane and desflurane anasthetic agents under low flow (one litre/min) conditi | Duration of surgery 4hours,4-6 hours, more than 6hours
  To compare the mac hour consumption of sevoflurane anasthetic agents under low flow (one litre/min) conditions To calculate the carbon foot print of sevoflurane and desflurane in the low flow anaesthesia being used in this study
To calculate the carbon foot print of sevoflurane and desflurane in low flow anaesthesia | Duration of surgery
  Carbon foot print calculation according to the formula

SECONDARY OUTCOMES:
To test whether significant generation of carbon monoxide occurs due to interaction of sevoflurane / desflurane with sodalime in the closed circuit. | end of surgery
  To test whether significant generation of carbon monoxide occurs due to interaction of sevoflurane / desflurane with sodalime in the closed circuit.

CONTACTS AND LOCATIONS:
Locations (1):
- RGCI& RC, Delhi, India

IPD SHARING:
Plan to Share IPD: No